CLINICAL TRIAL: NCT07284797
Title: A Phase 1, First-in-Human, Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of XmAb657 in Healthy Participants and in Participants With Idiopathic Inflammatory Myopathy
Brief Title: A Phase 1 Open-label Study to Evaluate Safety in Healthy Participants and Participants With Idiopathic Inflammatory Myopathy (IIM)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb657-01
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Idiopathic Inflammatory Myopathies
Keywords: Myopathy; Myositis
MeSH Terms: conditions — Myositis; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): XmAb657 administered SC
  Interventions: Biological: XmAb13676

INTERVENTIONS:
Biological: XmAb13676 — Biological

SUMMARY:
The purpose of this study is to determine the safety and tolerability of XmAb657 in healthy participants and participants with IIM. Participants will be given XmAb657 subcutaneously (SC) by injection under the skin.

DETAILED DESCRIPTION:
This is a Phase 1 study to determine the safety, tolerability, pharmacokinetic (PK), and pharmacodynamics (PD), and immunogenicity of XmAb657 in healthy adult participants and participants with IIM.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants - Adult participants in good health

Idiopathic inflammatory myopathy participants - Adult participants that meet the 2017 European Alliance of Association Rheumatology (EULAR)/American College of Rheumatology (ACR) classification of Idiopathic inflammatory myopathy

Idiopathic inflammatory myopathy participants - Stable doses of Idiopathic inflammatory myopathy medications prior to screening

All participants - Use of highly effective methods of contraception

Exclusion Criteria:

* Major surgery within 12 weeks prior to screening or planned within 12 months after dosing
* Recurrent infections or active clinically significant infection
* Active or untreated latent tuberculosis
* Cancer or history of cancer or lymphoproliferative disease within the previous 5 years
* Uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease

Note: Additional, more specific inclusion/exclusion criteria are defined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Through Week 24

SECONDARY OUTCOMES:
Serum concentration of XmAb657 | Through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Mark Osterman, MD, MSCE, Study Director — Xencor, Inc.
Locations (1):
- Xencor Investigative Site, Melbourne, Australia